CLINICAL TRIAL: NCT02549963
Title: A Prospective, Multi-Center, Pilot Study to Compare the Safety and Effectiveness of WATCHMAN Left Atrial Appendage Occlusion Device With Rivaroxaban for Stroke Prevention in Patients With Atrial Fibrillation
Brief Title: Evaluation of WATCHMAN Left Atrial Appendage Occlusion Device in Patients With Atrial Fibrillation Versus Rivaroxaban
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shulin Wu (Other)
Collaborators: Wuhan Asia Heart Hospital (Other); Beijing Anzhen Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Medical College (Other); First Affiliated Hospital of Jinan University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor-Investigator, Shulin Wu, Director of Guangdong Cardiovascular Institute, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GDCI 201501
Record Dates: First submitted 2015-09-08; First posted 2015-09-15 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WATCHMAN LAA Occlusion Device (Experimental): Subjects assigned to receive the WATCHMAN Left Atrial Appendage Occlusion Device.
  Interventions: Device: WATCHMAN Left Atrial Appendage Occlusion Device
- Rivaroxaban (Active Comparator): Subjects assigned to receive the Rivaroxaban therapy.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Device: WATCHMAN Left Atrial Appendage Occlusion Device
  Other Names: WATCHMAN Left Atrial Appendage Closure
  Arms: WATCHMAN LAA Occlusion Device
Drug: Rivaroxaban
  Other Names: Novel Oral Anticoagulant
  Arms: Rivaroxaban

SUMMARY:
This is a prospective, multi-center, randomized, pilot study comparing the WATCHMAN left atrial appendage occlusion device with Rivaroxaban therapy in patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal, persistent or permanent non-valvular atrial fibrillation
* Eligible for LAAO and long-term rivaroxaban therapy
* Calculated CHA2DS2-VASc score of 2 or greater.

Exclusion Criteria:

* Contraindicated/allergic to aspirin, clopidogrel and novel oral anticoagulants.
* Indicated for clopidogrel therapy or has taken clopidogrel within 7 days prior to enrollment.
* History of atrial septal repair or has an atrial septal defect/patent foramen ovale device.
* History of valvular heart disease.
* Implanted mechanical valve prosthesis.
* New York Heart Association Class IV congestive heart failure or left ventricular ejection fraction less than 30%.
* Patient has left atrial/left atrial appendage thrombus screened by echocardiography
* Platelet<100*109/L or hemoglobin<100g/L
* Expected lifespan less than 1 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint | 2 year
  All Stroke or Systemic embolism or Cardiovascular death

SECONDARY OUTCOMES:
All bleeding event | 2 year
  Any bleeding with a need for hospitalization, instrumental procedure or discontinuation of anticoagulation or antithrombotic treatment.
Major bleeding event | 2 year
  An overt bleeding accompanied by one or more of the following: a decrease in hemoglobin level of 20 g/l or more over a 24-hour period, transfusion of 2 or more units of packed red cells, bleeding at a critical site (intracranial, intraspinal, intraocular, pericardial, intramuscular with compartment syndrome, or retroperitoneal), or fatal bleeding
Technical and procedure related event | 45 days
  A pericardial effusion with a need for drainage, surgical or pericardiocentesis, or cardioembolic event during the procedure, or significant periprocedural bleeding (i.e. major vascular bleeding with a need for surgical revision, or blood concentrate transfusion), or device embolization, or thrombus of the device with a consequent cardioembolic event.
Cognitive function change | 2 year
  Montreal Cognitive Assessment(MoCA) will be performed to detect cognitive function change.The differences between the MoCA test score in WATCHMAN group and in a control group of Rivaroxaban

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - The first Affiliated Hospital of Guangzhou medical University, Guangzhou, Guangdong
  - The first affiliated hospital of Jinan university, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The second Affiliated Hospital of Guangzhou medical University, Guangzhou, Guangdong
  - Guangdong Cardiovascular Institute, Guangdong General Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong
  - Wuhan Asia Heart Hospital, Wuhan, Hubei

REFERENCES:
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957